CLINICAL TRIAL: NCT01608789
Title: Virtue® Male Sling European Study
Brief Title: Virtue® European Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU012
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Stress Urinary Incontinence
Keywords: Male sling; Stress Urinary Incontinence; Urination Disorders; Urologic Diseases
MeSH Terms: conditions — Urinary Incontinence, Stress; Urination Disorders; Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Virtue® Male Sling (Experimental): Patient implanted Virtue® Male Sling
  Interventions: Device: Virtue® Male Sling

INTERVENTIONS:
Device: Virtue® Male Sling — The Coloplast Virtue® Male Sling is a Class II, implantable, sub-urethral, permanent, non-absorbable support sling indicated for the surgical treatment of male stress urinary incontinence (SUI) resulting from intrinsic sphincter deficiency (ISD).

SUMMARY:
This study is a prospective, single arm, non-randomized, multi-center clinical study that will be conducted in Europe. It is designed to assess efficacy and safety of the Virtue® Male Sling in post-prostatectomy urinary incontinence.

DETAILED DESCRIPTION:
This study is a prospective, single arm, non-randomized, multi-center clinical study that will be conducted at up to thirteen centers in Europe. It is designed to assess efficacy and safety of the Virtue® Male Sling. One hundred and twenty-one subjects, satisfying criteria for selection, will be implanted with no more than 15 implanted per site. The study's primary end point will be evaluated at 12 months with continued data collection through 36 months.

ELIGIBILITY:
Inclusion Criteria:

* The subject has an estimated life expectancy of more than 5 years

  * The subject has confirmed stress urinary incontinence (SUI) through medical history, urodynamics, and/or physical exam for at least 6 months
  * The subject has intrinsic sphincter deficiency due to radical prostatectomy completed at least 1 year prior to implantation date
  * The subject has a good bladder function
  * The subject has failed non-invasive therapies, eg. Pelvic Floor/Kegel exercises, behavioral modification, or biofeedback, for at least 6 months
  * The subject is willing to have the Virtue® Male Sling implanted
  * The subject is able and willing to complete all follow-up visits and procedures indicated in this protocol

Exclusion Criteria:

* The subject is unable or unwilling to comply with all follow-up requirements according to the study protocol

  * The subject has an active urinary tract infection or active skin infection in region of surgery (temporary exclusion)
  * The subject has compromised immune systems or any other conditions that affect healing
  * The subject has serious bleeding disorders
  * The subject has an urinary incontinence that is not mainly a stress urinary incontinence
  * The subject has a stress urinary incontinence due to TransUrethral Resection or laser surgery of the Prostate (TURP)
  * The subject has incontinence due to neurogenic causes defined as multiple sclerosis, spinal cord/brain injury, CVA, detrusor-external sphincter dyssynergia, Parkinson's disease, or similar conditions
  * The subject had a previous implant (male sling, Artificial Urinary Sphincter) to treat stress urinary incontinence (previous implanted bulking agents are allowed)
  * The subject has undergone radiation, cryosurgery, or brachy therapy to treat prostate or other pelvic cancer within 6 months
  * The subject is likely to undergo radiation therapy within the next 3 months
  * The subject has a postvoid residual (PVR) > or = 150mL
  * The subject has recently required transurethral instrumentation for urethral or urethro-vesical anatomosis stricture within the previous 6 months
  * The subject is enrolled in a concurrent clinical study of any treatment (drug or device) that could affect continence function without the sponsors' approval
  * The subject is deemed unfit for male sling implantation or participation in a research protocol as determined by the attending physician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-08-27 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Improvement of urinary incontinence based on 24-hour pad test | 1 year
  The primary effectiveness end point will be improvement in pad weight defined as at least a 50% reduction in 24-hour pad weight from baseline to 12-months.
Safety of the device characterized by reported adverse events | 1 year
  Safety of the device, including the implant procedure.

SECONDARY OUTCOMES:
Improvement of urinary incontinence based on 24-hour pad test | Baseline, 1 month, 3 months, 6 months, 2 years, 3 years
  24 hour pad weight tests will be administered at baseline, 1, 3, 6, 12, 24 and 36 months and the difference reported. Outcomes reported will include mean paired change from baseline as well as the proportion or patients improving by at least 50% from baseline
Improvement of urinary incontinence based on number of pad used | baseline,1 month, 3 months, 6 months, 1 year, 2 years and 3 years
  Number and types of pads used will be collected at baseline,1, 3, 6, 12, 24 and 36 months and the difference reported.
Improvement of urinary incontinence based on PGI-I | 1 month, 3 months, 6 months, 1 year, 2 years, 3 years
  Patient global Impression of improvement
Assessment of the frequency, severity and impact on quality of life of urinary incontinence based on ICIQ-UI short form | baseline, 1 months, 3 months, 6 months, 1 year, 2 years and 3 years
  Base on International Consultation on Incontinence questionnaire-Urinary Incontinence short-form
Patient satisfaction questionaire | 1 month, 3 months, 6 months, 1 year, 2 years, 3 years
  the patient reported level of satisfaction in implantation sling procedure.
Safety of the device characterized by reported adverse events | Intraoperative, 1 month, 3 months, 6 months, 2 years, 3 years
  Safety of the device, including the implant procedure.

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (2):
  - Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- France (3):
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Groupe Hospitalo Universitaire Carémeau, Nîmes
  - Hôpital de la Pitié-Salpêtrière, Paris
- Germany (2):
  - Heilig Geist Krankenhaus, Cologne
  - Universitätsklinikum Schleswig-Holstein, Kiel
- Mater Private Hospital, Dublin, Ireland
- Italy (2):
  - Istituto europeo di Oncologia, Milan
  - Hospital Santa Maria della Misericordia, Udine
- Leiden University Medical Center, Leiden, Netherlands
- Spain (2):
  - Fundacio Puigvert - Universitat Autonoma de Barcelona, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No